CLINICAL TRIAL: NCT05104580
Title: PrOgnostic Implications of PRe-stent Pullback Pressure GradIent and Post-stent Quantitative Flow Ratio in Patients UnderGoing Percutaneous Coronary INtervention
Acronym: CHART-ORIGIN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-20211021
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: High pre-PCI PPG index and high post-PCI QFR
  Interventions: Device: Quantitative Flow Ratio derived PPG
- Group 2: Low pre-PCI PPG index and high post-PCI QFR
  Interventions: Device: Quantitative Flow Ratio derived PPG
- Group 3: Low post-PCI QFR regardless of pre-PCI PPG index
  Interventions: Device: Quantitative Flow Ratio derived PPG

INTERVENTIONS:
Device: Quantitative Flow Ratio derived PPG — From coronary angiographic images, QFR will be calculated and virtual pullback curve will be abstracted and PPG index will be calculated as:
  PPG index={MaxPPG20mm/△QFRvessel+(1-length with functional disease/Total vessel length) }/2.

SUMMARY:
The purpose of this study is to investigate the prognostic implication of pre-percutaneous coronary intervention (PCI) focal or diffuse disease patterns combined with post-PCI quantitative flow ratio (QFR).

DETAILED DESCRIPTION:
Coronary diffuse disease associates with poor outcomes, but little is known about whether this prognostic value retains after PCI, especially in those with good post-PCI physiologic results.

QFR can provide the virtual pullback curve by depicting pressure at each point along the interrogated vessel, which can be used to calculate the pullback pressure gradient (PPG) index, this index has been shown to be able to suggest the physiological plaque distribution and to discriminate focal from diffuse disease. Absolute quantification of coronary diffuseness makes it possible to evaluate the prognostic value of baseline coronary diffuseness before stent implantation, which is rarely investigated till now.

The CHART-ORIGIN study aims to investigate the independent and additive prognostic implications of pre-PCI functional disease patterns assessed by PPG with post-PCI QFR in vessels with stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one vessel with measurable QFR
* PPG index can be calculated from virtual QFR pullback curve;
* The patient is willing to comply with specified follow-up evaluations;
* Patients who agree to accept the follow-up visits.

Exclusion Criteria:

* Culprit vessels for ACS myocardial infarction;
* Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure;
* Patient has other medical illness (e.g., cancer, known malignancy, congestive heart failure, organ transplant recipient or candidate) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than 1 year);
* Patient has a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel/ticlopidine, stainless steel alloy, cobalt chromium, rapamycin, styrene-butylenes-styrene or poly-lactic acid (PLA) polymer, and/or contrast sensitivity that cannot be adequately pre-medicated;
* Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study;
* Currently participating in another investigational drug or device study or patient in inclusion in another investigational drug or device study during follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1,395 patients with 1,685 target vessels with measurable QFR and PPG index from the PANDA-III study (Comparison of BuMA eG Based BioDegradable Polymer Stent With EXCEL Biodegradable Polymer Sirolimus-eluting Stent in "Real-World" Practice) (NCT02017275).
Sampling Method: Non-Probability Sample
Enrollment: 1395 (Estimated)
Dates: Start 2021-10-30 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Vessel-oriented composite outcome | at 2 years from index procedure
  Vessel-oriented composite outcome (VOCO) including vessel related ischemia-driven target vessel revascularization, vessel-related myocardial infarction (MI), and cardiac death.

SECONDARY OUTCOMES:
Cardiac death or vessel-related MI | at 2 years from index procedure
  Cardiac death or vessel-related MI
Vessel-related MI | at 2 years from index procedure
  Vessel-related MI
Cardiac death | at 2 years from index procedure
  Cardiac death
Ischemia-driven target vessel revascularization | at 2 years from index procedure
  Ischemia-driven target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Professor, Study Chair — Fudan University; Bo Xu, MBBS, Principal Investigator — Fu Wai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xu B, Gao R, Yang Y, Cao X, Qin L, Li Y, Li Z, Li X, Lin H, Guo Y, Ma Y, Wang J, Nie S, Xu L, Cao E, Guan C, Stone GW; PANDA III Investigators. Biodegradable Polymer-Based Sirolimus-Eluting Stents With Differing Elution and Absorption Kinetics: The PANDA III Trial. J Am Coll Cardiol. 2016 May 17;67(19):2249-2258. doi: 10.1016/j.jacc.2016.03.475. PMID 27173037
- [Background] Dai N, Hwang D, Lee JM, Zhang J, Jeon KH, Paeng JC, Cheon GJ, Koo BK, Ge J. Feasibility of Quantitative Flow Ratio-Derived Pullback Pressure Gradient Index and Its Impact on Diagnostic Performance. JACC Cardiovasc Interv. 2021 Feb 8;14(3):353-355. doi: 10.1016/j.jcin.2020.10.036. No abstract available. PMID 33541549
- [Background] Dai N, Zhang R, Hu N, Guan C, Zou T, Qiao Z, Zhang M, Duan S, Xie L, Dou K, Zhang Y, Xu B, Ge J. Integrated coronary disease burden and patterns to discriminate vessels benefiting from percutaneous coronary intervention. Catheter Cardiovasc Interv. 2022 Jan 1;99(1):E12-E21. doi: 10.1002/ccd.29983. Epub 2021 Oct 15. PMID 34652068
- [Derived] Dai N, Yuan S, Dou K, Zhang R, Hu N, He J, Guan C, Zou T, Qiao Z, Duan S, Xie L, Yu Y, Zhang Y, Xu B, Ge J. Prognostic Implications of Prestent Pullback Pressure Gradient and Poststent Quantitative Flow Ratio in Patients Undergoing Percutaneous Coronary Intervention. J Am Heart Assoc. 2022 Jun 7;11(11):e024903. doi: 10.1161/JAHA.121.024903. Epub 2022 Jun 3. PMID 35656982